CLINICAL TRIAL: NCT00204789
Title: Phase 2b Difluoromethylornithine (DFMO) Chemoprevention of Skin Cancer in Organ Transplant Recipients (OTR)
Brief Title: Difluoromethylornithine (DFMO) Chemoprevention of Skin Cancer in Organ Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2001-414; CO00318
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2007-12

CONDITIONS: Post-solid Organ Transplant; Skin Neoplasms
MeSH Terms: conditions — Skin Neoplasms | interventions — Eflornithine

INTERVENTIONS:
Drug: Difluoromethylornithine

SUMMARY:
This is a double blind, placebo controlled study of 52 patients who are at least one-year post-solid organ transplant. Subjects will receive either 12 months of DFMO or a placebo. The specific aims are to determine if DFMO at 500 mg daily will be well tolerated for 12 months and not affect organ transplant viability; will inhibit 12-O-tetradecanoylphorbol-13-acetate (TPA)-induced ornithine decarboxylase (ODC) in skin biopsies by approximately 50% for the 12 months of therapy; and will be able to decrease polyamine levels in skin biopsies for the 12 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* >1 year post-solid organ transplant of kidney, liver, pancreas, pancreas/kidney
* Adequate organ function
* Hearing age/gender appropriate
* At high risk for developing skin cancer
* Immunosuppressant levels and doses show stable graft function

Exclusion Criteria:

* Use of concomitant Retin-A, Efudex, Accutane or psoralen and ultraviolet light A (PUVA)
* Systemic therapy for cancer treatment or prophylaxis
* Use of concomitant azathioprine, antiseizure medications, non-steroidal anti-inflammatory drugs [NSAIDs] (other than cardioprotective doses of aspirin)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2003-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To determine if DFMO at 500 mg daily will be well tolerated and not affect organ transplant viability | for 12 months

SECONDARY OUTCOMES:
To determine if DFMO will inhibit TPA-induced ODC in skin biopsies by approximately 50% | for the 12 months of therapy
To determine if DFMO will be able to decrease polyamine levels in skin biopsies | for the 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Howard H Bailey, MD, Principal Investigator — University of Wisconsin, Madison